CLINICAL TRIAL: NCT03730571
Title: Prospective, Multi-center, Non-Randomized Controlled Trial of Vascular Closure Using the AbsorbaSeal 6 French Vascular Closure Device
Brief Title: The AbsorbaSeal Vascular Closure Device Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient closure
Sponsor: ID3 Medical (Other)
Collaborators: CyndRx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CP002CE
Record Dates: First submitted 2018-09-28; First posted 2018-11-05 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AbsorbaSeal 6Fr Vascular Closure Device (Experimental): Patients whose access site will be closed with the AbsorbaSeal 6Fr Vascular Closure Device
  Interventions: Device: AbsorbaSeal 6Fr Vascular Closure Device

INTERVENTIONS:
Device: AbsorbaSeal 6Fr Vascular Closure Device — Patients whose access site will be closed with the AbsorbaSeal 6Fr Vascular Closure Device

SUMMARY:
This study investigates the efficacy and safety of the AbsorbaSeal 6Fr Vascular Closure device (VCD) for the closure of access site of patients requiring percutaneous diagnostic or interventional procedures. An expected total of 50 patients will be enrolled in this study. A total of 12 patients (4 patients per site) will be treated as roll-in phase, prior to enrollment of the first patient. The primary objective of this study is to assess the safety and effectiveness of the AbsorbaSeal 6Fr VCD. Enrollment into this study will include anatomically eligible patients requiring diagnostic and interventional procedures. Following physician training, patients will be enrolled. Efficacy and safety analyses will be based on these patients.Patients will be followed procedurally to discharge, at one month, (follow-up commitment). Secondary objectives are to further characterize adverse events (serious and non-serious), clinical utility measures and health-related quality of life.

DETAILED DESCRIPTION:
With the increased number of percutaneous interventions being performed in outpatient settings there is a growing need to obtain faster, safer, and more secure hemostasis following these outpatient procedures. CyndRx believes an improved VCD will lead to more widespread use and ultimately improve patient outcomes. The AbsorbaSeal Vascular Closure Device (ABS-6) has been developed to meet this need. The ease of use and automatic deployment of the device will eliminate the learning curve associated with the use of VCDs. The active closure system used in the ABS-6 ensures a secure closure with every deployment. The composition of the seal used is completely bio-absorbable and does not require the use of adjunct materials (i.e. collagen, sutures, staples, etc.) needed in many of the devices currently available.

The First In Man (FIM) trial demonstrated the safety and efficacy of the ABS-6 system in humans (N=20). To further evaluate the safety and efficacy, up to 50 patients will be enrolled in the CP002CE-study.

The primary objective of this study is to assess the safety and effectiveness of the AbsorbaSeal 6Fr VCD. Enrollment into this study will include anatomically eligible patients requiring diagnostic and interventional procedures. Patients will be followed procedurally to discharge, at one month, (follow-up commitment). Secondary objectives are to further characterize adverse events (serious and non-serious), clinical utility measures, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 85 years of age
* Male and Female
* Patient/legal representative provides written informed consent
* Patient is scheduled for a coronary or peripheral diagnostic or interventional procedure
* Patient is able to undergo emergent vascular surgery if a complication related to the VCD necessitates such surgery
* Patient has a 6 french arterial puncture located in the common femoral artery
* Target vessel has a lumen diameter ≥ 5 mm
* Patient is willing and able to complete follow-up
* Catheterization procedure is planned and elective

Exclusion Criteria:

* Prior target artery closure with any closure device or closure with manual compression ≤ 30 days prior to the cardiac or peripheral catheterization procedure
* Patients with a history of significant bleeding or with any known or documented bleeding disorders, such as Thrombocytopenia (with < 100,000 platelet count), Von Willebrand's disease, anemia (Hgb < 10 g/dL, Hct < 30%), thrombasthenia, decreased fibrinogen (< 200 mg/dL), and Factor V deficiency
* Acute ST-elevation myocardial infarction ≤ 48 hours prior to the cardiac or peripheral catheterization procedure
* Patient is ineligible for in-lab catheterization lab introducer sheath removal
* Concurrent participation in another investigational device or drug trial
* Thrombolytic therapy (e.g. streptokinase, urokinase, t-PA) ≤ 24 hours prior to the cardiac or peripheral catheterization procedure
* Evidence of a preexisting hematoma, arteriovenous fistula, or pseudoaneurysm at the access site prior to start of femoral artery closure procedure
* Prior femoral vascular surgery or vascular graft in region of access site or contralateral common femoral artery
* The targeted femoral artery is tortuous or requires a sheath length > 10 cm
* Patient is pregnant or breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Treatment success | 30 days post-index procedure
  Composite of (1) procedural technical success (successful vascular access and ABS-6 delivery, deployment and catheter removal), (2) absence of vascular complications (arteriovenous fistula, femoral neuropathy, hematoma >6cm, hemorrhage, infection, lymphocele, thrombosis/occlusion/distal emboli/stenosis, vascular injury) (3) absence of major adverse events (all-cause death, cardiac morbidity, neurological complications, renal failure, respiratory complications, secondary intervention for groin complications)

SECONDARY OUTCOMES:
Number of Adverse events | 30 days post-index procedure
  All adverse events will be monitored. A serious adverse event is defined as an event that results in death, is life threatening, requires inpatient hospitalization or that prolongs hospitalization, results in persistent or significant disability/incapacity
Volume of contrast media used during index procedure | Intraoperative
  Volume of contrast media used (ml)
Fluoroscopy time during index procedure | Intraoperative
  Fluoroscopy time (min)
Estimated blood loss during index procedure | Intraoperative
  Estimated blood loss (ml)
Time to hemostasis after index procedure | Intraoperative
  Time to hemostasis (min)
Total procedure time of index procedure | Intraoperative
  Total procedure time (min)
Anesthesia time of index procedure | Intraoperative
  Anesthesia time (min)
Total time of initial hospitalization stay | Up to 1 month post-index procedure
  Total time of initial hospitalization stay (h:min)
Analgesic usage after index-procedure | 1-day post-index procedure
  Arterial access site pain-related analgesic usage after index procedure until patient discharge
Pain Evaluation | 1-day post-index procedure and 1 month follow-up
  Self-reported groin pain scale (0 (no pain) - 10 (excessive pain))

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Principal Investigator — ID3 Medical
Locations (3):
- Belgium (3):
  - O.L.V. Hospital, Aalst
  - Imelda Hospital, Bonheiden
  - A.Z. Sint-Blasius, Dendermonde